CLINICAL TRIAL: NCT00850083
Title: Accuracy of Measurement of Surface Body Temperature Using the Health e Pod Device (Card Guard) Compared to Gold Standard Equipment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Eran Kozer, Assaf Harofeh Medical Center
Other Study IDs: 152/08
Record Dates: First submitted 2009-02-23; First posted 2009-02-24 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: All Children Admitted to the ED; Children With Fever
Keywords: Fever; Children
MeSH Terms: conditions — Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children in the ED

SUMMARY:
Objective To evaluate the accuracy of data acquisition by Health e pod device in measurement of body temperature, to compare it to a standard body temperature measure equipment About 400 consecutive patients admitted to PEU in Assaf Harofeh Medical Center will compile the Study Population.

Basic vital signs will be recorded on admission and during hospitalization as per the PEU policy and not in particular for this study.

As a part of routine check-up all admitted patients undergo body temperature measure (oral or rectal - as per the PEU policy and with PEU devices).

Following an explanation and patient agreement, eligible patients (and their legal guardian) will sign informed consent and enter the study. The health e pod device will be applied to measure body temperature, immediately after the standard temperature measure has been performed by the PEU professional.

ELIGIBILITY:
Inclusion Criteria:

* Signed an Informed Consent by the patients' legal custodian / guardian (and assent by the patient when applicable).
* Age 0 to 18 years
* Clinically stable patients hospitalized in PEU.

Exclusion Criteria:

* Implanted pacemaker or defibrillator.
* Patients participating in other clinical trail.

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children visiting the pediatric emergency unit
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2009-03; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Agreament between measurments by Health e pod device and the gold standard reference device. | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel